CLINICAL TRIAL: NCT04107558
Title: Healthy Volunteer Undergoing Painful Stimuli With and Without Virtual Reality Hypnosis (VRH)
Brief Title: Healthy Volunteer Undergoing Painful Stimuli With and Without Hypnosis and Virtual Reality
Acronym: SMARTHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oncomfort (Industry)
Collaborators: University of Liege (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pilot 1
Record Dates: First submitted 2019-09-23; First posted 2019-09-27 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Digital Sedation
Keywords: Virtual reality , hypnosis, pain, anxiety, anesthesia
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will undergo painful stimuli without HVR followed by a session with HVR. Subjects are their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painful stimuli with Hypnosis and Virtual Reality (Experimental): After 5 minutes of rest, we start with painful stimuli during 10 minutes. This session takes place under hypnosis
  Interventions: Device: Virtual Reality
- Painful stimuli without Hypnosis and Virtual reality (No Intervention): After 5 minutes of rest, we start with painful stimuli during 10 minutes.

INTERVENTIONS:
Device: Virtual Reality — Subjects will undergo painful stimuli without HVR followed by a session with HVR. Subjects are their own control
  Arms: Painful stimuli with Hypnosis and Virtual Reality

SUMMARY:
The main purposes of this study are as follows:

Compare the effect of painful stimuli with and without Hypnosis and Virtual Reality (HVR) on healthy volunteers.

* Use of sensors and captors to monitor physiological and neurophysiological changes by painful stimulus
* Monitor level of pain and anxiety with and without HVR
* Monitor level of unpleasantness of the pain with and without HVR
* Monitor level of Anxiety, Absorption, Dissociation, Satisfaction and Comfort with and without HVR

DETAILED DESCRIPTION:
The control of pain and anxiety in a hospital environment is usually managed by pharmacological means that involve a series of risks and side effects.

For many years, non-drug solutions have been of interest to the public and the care staff. The benefits of hypnosis and of virtual reality are highlighted in many studies and today allow a different approach to medicine. It is important to invest in tools that are less expensive and also effective for the well-being of the patient and the care staff. The use of a blended solution using both clinical hypnosis and virtual reality has been only scarcely documented.

ELIGIBILITY:
Inclusion Criteria:

- 18 years old to 70 years of age

Exclusion Criteria:

* Deaf subject
* Blind
* Non-proficiency in French (research language)
* Psychiatric disorder
* Patient under 18 years old
* Phobia of deep water
* Head or face wounds
* Claustrophobia
* Neurological disease
* Allergy to cutaneous electrodes
* Chronic pain and/or chronic analgesics consumption
* Medication affecting the autonomic nervous system
* Dizziness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Compare physiological and neurophysiological changes to painful stimulation with and without Hypnosis and Virtual Reality (HVR) | During the procedure
  To understand the effect of VRH on the Physiological and neurophysiological parameters recorded by sensors and captors

SECONDARY OUTCOMES:
Pain and anxiety | Immediately before and after the procedure
  To understand the effect of VRH on the level of pain and anxiety. Pain and anxiety Pain assessed by visual analogue scale (VAS).
  Participants will record their pain intensity rating on a Visual analogue scale where 0 = No pain and 10 = worst imaginable pain. Subject will record also their level of anxiety on the same VAS
Unpleasantness of the pain | Immediately after the procedure
  To understand the effect of VRH on the level of the unpleasantness of the pain assessed by visual analogue scale. Participants similarly record their pain unpleasantness parting on a VAS where 0= not at all unpleasant and 10= most unpleasantness imaginable.
Absorption, Dissociation, Satisfaction and comfort, presence and cybersickness | Immediately after the procedure
  To understand the effect of VRH on the level of Absorption, Presence, Dissociation, Satisfaction and comfort assessed by visual analogue scale. Participant record their level of absorption, dissociation, satisfaction and comfort on a VAS where 0 = no absorption, no dissociation, no satisfaction and no comfort at all. 10 is the opposite

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Liège- CHU, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No